CLINICAL TRIAL: NCT03637790
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE STUDY TO ESTIMATE THE EFFECT OF REPEAT-DOSE RIFAMPIN ON THE PHARMACOKINETICS OF PF-04965842 IN HEALTHY SUBJECTS
Brief Title: Drug Interaction Study Evaluating the Effect of Rifampin on PK and Safety of PF 04965842.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: B7451019; 2018-002167-25 (EudraCT Number)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — abrocitinib; Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF 04965842 (Other): In Period 1, subjects will be administered a single oral 200 mg dose of PF 04965842 in the morning on Day 1 under fasted conditions.
  Interventions: Drug: PF-04965842
- Rifampin and PF 04965842 (Other): In Period 2, subjects will receive rifampin 600 mg QD in the mornings of Day 1 to Day 7, approximately 1 hour before the morning meal. On the morning of Day 8, after an overnight fast of approximately 9 hours, subjects will be administered rifampin 600 mg 1 hour prior to administration of a single 200 mg oral dose of PF 04965842.
  Interventions: Drug: PF-04965842; Other: rifampin

INTERVENTIONS:
Drug: PF-04965842 — single oral 200 mg dose of PF 04965842 in the morning on Day 1 under fasted conditions.In Period 2, subjects will receive rifampin 600 mg QD in the mornings of Day 1 to Day 7, approximately 1 hour before the morning meal. On the morning of Day 8, after an overnight fast of approximately 9 hours, subjects will be administered rifampin 600 mg 1 hour prior to administration of a single 200 mg oral dose of PF 04965842.
Other: rifampin — In Period 2, subjects will receive rifampin 600 mg QD in the mornings of Day 1 to Day 7, approximately 1 hour before the morning meal. On the morning of Day 8, after an overnight fast of approximately 9 hours, subjects will be administered rifampin 600 mg 1 hour prior to administration of a single 200 mg oral dose of PF 04965842
  Arms: Rifampin and PF 04965842

SUMMARY:
This is a Phase 1 open label, 2 period, single fixed sequence study designed to evaluate the effect of repeat dose oral rifampin on single dose PF 04965842 PK after a single 200 mg oral dose in healthy subjects. A total of 12 healthy male and/or female subjects will be enrolled in the study so that at least 10 subjects will complete the study.

Subject will report to the clinical research unit (CRU) at least 12 hours prior to Day 1 dosing in Period 1 and will be required to stay in the CRU for 11 days and 10 nights. Genotyping samples for CYP2C19 and CYP2C9 will be collected predose in Period 1 only. In Period 1, subjects will be administered a single oral 200 mg dose of PF 04965842 in the morning on Day 1 under fasted conditions. No food will be allowed for at least 4 hours postdose and undergo serial blood sample collection for 24 hours postdose to characterize the PK profile of PF 04965842.

In Period 2, subjects will receive rifampin 600 mg QD in the mornings of Day 1 to Day 7, approximately 1 hour before the morning meal. On the morning of Day 8, after an overnight fast of approximately 9 hours, subjects will be administered rifampin 600 mg 1 hour prior to administration of a single 200 mg oral dose of PF 04965842. Subjects will remain in a fasted state for 4 hours after dosing with PF 04965842 and undergo serial blood sample collection for 24 hours post PF 04965842 dosing to characterize the PK profile of PF 04965842. Subjects will be discharged from the CRU on Day 9 of Period 2 after all study procedures are completed. The subject will be required to return to the CRU for on site follow up visits 7 14 days, and have a follow up phone contact 28 35 days after the last dose of PF 04965842.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. Healthy female subjects and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12 lead ECG, or clinical laboratory tests.

   Female subjects of non childbearing potential must meet at least 1 of the following criteria:
   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.
2. Body mass index (BMI) of 17.5 to 30.5 kg/m2 and a total body weight >50 kg (110 lb).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing). Evidence of acute exacerbation of dermatological condition (eg, AD, eczema or psoriasis) or visible rash present during physical examination. Subjects with history of psoriasis, AD or eczema can be included in the study.
2. Subjects, who according to the product label for rifampin, would be at increased risk if dosed with rifampin.
3. Any condition possibly affecting drug absorption (eg, gastrectomy).
4. A positive urine drug test.
5. History of regular alcohol consumption exceeding 14 drinks/week for female subjects or 21 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
6. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
7. Screening supine systolic BP <90 mm Hg or >140 mm Hg following at least 5 minutes of supine rest OR Screening supine diastolic BP <50 mm Hg or >90 mm Hg following at least 5 minutes of supine rest.

   If a subject meets any of these criteria, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
8. Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
9. Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use 1 highly effective method of contraception as outlined in this protocol Contraception section for the duration of the study and for at least 28 days after the last dose of investigational product.
10. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level 1.5 × upper limit of normal (ULN);
    * Total bilirubin level 1 × ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ULN.
11. Use of CYP2C19 inhibitors (eg, fluconazole, fluoxetine, fluvoxamine, ticlopidine omeprazole, voriconazole, cimetidine, esomeprazole, and felbamate) or inducers (eg, rifampin, ritonavir, efavirenz, enzalutamide, phenytoin, and St. John's Wort) within 28 days or 5 half lives (whichever is longer) prior to dosing.
12. Use of CYP2C9 inhibitors (eg, amiodarone, felbamate, fluconazole, miconazole, piperine, diosmin, disulfiram, fluvastatin, fluvoxamine, voriconazole, efavirenz, isoniazid) or inducers (eg, aprepitant, carbamazepine, enzalutamide, rifampin, ritonavir, nevirapine, phenobarbital, and St. John's Wort) within 28 days or 5 half lives (whichever is longer) prior to dosing.
13. Use of CYP3A4 inhibitors (eg, ketoconazole, ciprofloxacin, diltiazem) or other inducers (eg, phenytoin, carbamazepine) within 28 days or 5 half lives (whichever is longer) prior to dosing.
14. Known relevant history of elevated liver function tests (LFTs) or impaired liver function.
15. History of active or latent or inadequately treated tuberculosis (TB) infection, or a positive QuantiFERON TB Gold test.
16. Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of screening.

    * History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.
    * History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or considered clinically significant by the investigator within 6 months prior to screening.
17. History of receiving a live vaccine within 6 weeks prior to the first dose of investigational product, or is expected to receive a live vaccine within 6 weeks after the last dose of investigational product.
18. Have a known immunodeficiency disorder or a first degree relative with a hereditary immunodeficiency.
19. History or evidence of any malignancies with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
20. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of < 1 g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.

    Herbal supplements and hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone releasing intrauterine devices [IUDs], vaginal ring, and postcoital contraceptive methods) and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of investigational product.
21. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
22. History of sensitivity to heparin or heparin induced thrombocytopenia.
23. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb). A positive hepatitis B surface antibody (HepBsAb) finding as a result of subject vaccination is permissible.
24. A current or past medical history of conditions associated with thrombocytopenia, coagulopathy or platelet dysfunction.
25. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
26. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
27. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
28. Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day or 2 chews of tobacco per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Plasma PF 04965842 Cmax PK | Day 1 on period 1 and Days 1, 8 and 9 on period 2
  Maximum observed plasma concentration for PF 04965842
AUCinf for PF 04965842 | Day 1 on period 1 and Days 1, 8 and 9 on period 2
  Area under the curve from time zero to extrapolated infinite time tor PF 04965842

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs). | Screening up to 28-35 days after the last dose of PF 04965842 in period 2
  Number of subjects with adverse events (AEs).
Number of subjects with laboratory tests findings of potential clinical importance | Screening up to 7-14 days after the last dose of PF 04965842 in period 2
  Number of subjects with laboratory tests findings of potential clinical importance
Number of subjects with clinically significant abnormal vital signs | Screening up to 7-14 days after the last dose of PF 04965842 in period 2
  Number of subjects with clinically significant abnormal vital signs
Number of subjects with clinically significant abnormal Electrocardiograms (ECGs) | Screening up to 7-14 days after the last dose of PF 04956842 in period 2.
  Number of subjects with clinically significant abnormal Electrocardiograms (ECGs).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang X, Dowty ME, Wouters A, Tatulych S, Connell CA, Le VH, Tripathy S, O'Gorman MT, Winton JA, Yin N, Valdez H, Malhotra BK. Assessment of the Effects of Inhibition or Induction of CYP2C19 and CYP2C9 Enzymes, or Inhibition of OAT3, on the Pharmacokinetics of Abrocitinib and Its Metabolites in Healthy Individuals. Eur J Drug Metab Pharmacokinet. 2022 May;47(3):419-429. doi: 10.1007/s13318-021-00745-6. Epub 2022 Feb 28. PMID 35226304
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451019